CLINICAL TRIAL: NCT04317781
Title: Tagraxofusp (SL-401) Therapy for Blastic Plasmacytoid Dendritic Cell Neoplasm (BPDCN) Patients Post-Autologous or Post-Allogeneic Hematopoietic Cell Transplantation
Brief Title: Tagraxofusp in Treating Patients With Blastic Plasmacytoid Dendritic Cell Neoplasm After Stem Cell Transplant
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The protocol was terminated early due to slow participant accrual and the sponsor not willing to provide the study drug.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0646; NCI-2019-03832 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0646 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-03-19; First posted 2020-03-23 (Actual); Results first posted 2024-07-16 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Blastic Plasmacytoid Dendritic Cell Neoplasm
MeSH Terms: conditions — Blastic Plasmacytoid Dendritic Cell Neoplasm | interventions — tagraxofusp

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (tagraxofusp-erzs) (Experimental): Within day 45 and 180 after stem cell transplant, patients receive tagraxofusp-erzs IV over 15 minutes on days 1-3 of cycles 1-4 and days 1-2 of subsequent cycles. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Tagraxofusp-erzs

INTERVENTIONS:
Biological: Tagraxofusp-erzs — Given IV
  Other Names: Diphtheria Toxin(388)-Interleukin-3 Fusion Protein; DT(388)-IL3 Fusion Protein; DT388IL3 fusion protein; Elzonris; IL3R-targeting Fusion Protein SL-401; SL-401; Tagraxofusp; Tagraxofusp ERZS

SUMMARY:
This phase II trial studies the side effects of tagraxofusp in treating patients with blastic plasmacytoid dendritic cell neoplasm after stem cell transplant. Tagraxofusp is a type of immunotoxin that is made by linking a protein called IL-3 to a toxic substance. Tagraxofusp may help find cancer cells that express IL-3 and kill them without harming normal cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety of tagraxofusp-erzs (tagraxofusp) in patients with blastic plasmacytoid dendritic cell neoplasm (BPDCN) after autologous (auto) or allogeneic (allo) hematopoietic cell transplantation (HCT).

SECONDARY OBJECTIVES:

I. To estimate progression-free survival (PFS) in patients with BPDCN receiving maintenance therapy with tagraxofusp after auto-HCT or allo-HCT.

II. To estimate the overall survival (OS) in patients with BPDCN receiving maintenance therapy with tagraxofusp after auto-HCT or allo-HCT.

OUTLINE:

Within day 45 and 180 after stem cell transplant, patients receive tagraxofusp-erzs intravenously (IV) over 15 minutes on days 1-3 of cycles 1-4 and days 1-2 of subsequent cycles. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will be aged >= 18 years. Pediatric patients age 2 years and older will be considered on a case by case basis.
* Diagnosis of blastic plasmacytoid dendritic cell neoplasm (BPDCN) according to World Health Organization (WHO) classification or confirmed by hematopathology
* The patients must be in partial response or better
* > 30 days post-transplant without active or chronic infections
* Karnofsky performance status >= 60%; Lansky >= 60
* Left ventricular ejection fraction (LVEF) >= institutional lower limit of normal by multigated acquisition (MUGA) scan or echocardiogram within 30 days of first protocol treatment
* Diffusion capacity of the lung for carbon monoxide (DLCO) > 40% of predicted value (corrected for hemoglobin) within 3 months of registration
* Forced expiratory volume in 1 second (FEV1) > 40% of predicted value within 3 months of registration
* Forced vital capacity (FVC) > 40% of predicted value within 3 months of registration
* Serum creatinine =< 1.5 mg/dL (133 mmol/L)
* Serum albumin >= 3.2 g/dL (or >= 32 g/L) without IV albumin within the previous 72 hours
* Bilirubin =< 1.5 x the upper limit of normal ([ULN] except patients with Gilbert syndrome in whom bilirubin level of > 1.5 x ULN will be allowed)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 times ULN
* Hemoglobin >= 8 g/dL with or without transfusion in the last 7 days
* Absolute neutrophil count (ANC) >= 1000 without granulocyte colony stimulating factor (GCSF) or granulocyte-macrophage colony-stimulating factor (GMCSF) in the last 2 weeks prior to screening
* Platelets >= 50,000micro/mL
* For allo-HCT, no >= grade 2 visceral (gut or liver) acute graft versus host disease (GVHD) and no >= grade 3 or any other acute GVHD (patients with chronic GVHD will be allowed at the discretion of the investigator)
* Patient agrees to use acceptable contraceptive methods for the duration of time in the study, and to continue to use acceptable contraceptive methods for 2 months after the last tagraxofusp infusion
* Woman of child bearing potential (WOCBP) with a negative serum or urine pregnancy test within 14 days of tagraxofusp treatment
* Patient or patient's legal representative, parent(s) or guardian able to sign informed consent
* The patient can adhere to the study visit schedule and other protocol requirements, including follow-up for survival assessment

Exclusion Criteria:

* The patient has persistent clinically significant non-hematologic toxicities >= grade 2 (excluding alopecia, nausea, and fatigue)
* Evidence of central nervous system (CNS) involvement
* Uncontrolled and active pulmonary disease
* Requirement for oxygen treatment
* Receiving chemotherapy, radiotherapy or other anti-cancer therapy within 14 days of first dose of study drug. There must be at least a 6-week interval from the last immunotherapy therapy
* Uncontrolled infection
* Human immunodeficiency virus (HIV)/hepatitis B and/or C
* Any history of invasive malignancy in the last 2 years excluding any malignancy such as cervical cancer or skin cancer (excluding melanoma) that is considered cured at the time of screening
* Pregnant or breast-feeding woman
* Patient has uncontrolled intercurrent illness or medical/psychiatric condition that would limit compliance with study requirements or that would in the investigator's opinion place the patient at an unacceptably high risk for toxicities
* Clinical significant cardiopulmonary disease including uncontrolled or New York Heart Association (NYHA) class 3 or 4 congestive heart failure, uncontrolled angina, uncontrolled hypertension, uncontrolled arrhythmia, myocardial infarction or stroke within 6 months of first protocol treatment or corrected QT (QTc) > 480 ms

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-03-27 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Qaiser Bashir, MS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Wang SY, Thomassen K, Kurch L, Opitz S, Franke GN, Bach E, Platzbecker U, Kayser S. Combination of Tagraxofusp and Azacitidine Is an Effective Option for Relapsed Blastic Plasmacytoid Dendritic Cell Neoplasm After Allogeneic Hematopoietic Stem-Cell Transplantation. Clin Lymphoma Myeloma Leuk. 2021 Jul;21(7):e579-e582. doi: 10.1016/j.clml.2021.02.008. Epub 2021 Mar 2. No abstract available. PMID 33795208
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were registered at MD Anderson Cancer Center
Period: Overall Study
Arm/Group | Treatment (Tagraxofusp-erzs)
Started | 3
Completed | 0
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Disease relapse | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Tagraxofusp-erzs)
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Received Planned Tagraxofusp Post Transplant
Description: Participants completed at least 75% of planned tagraxofusp doses in at least 4 cycles of therapy.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Tagraxofusp-erzs)
Number analyzed (Participants) | 3
Participants | 1

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Participant alive and disease free one year post transplant
Time Frame: From treatment start date to date of disease progression or death, assessed up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Tagraxofusp-erzs)
Number analyzed (Participants) | 3
Participants | 2

3. Secondary Outcome: Overall Survival (OS)
Description: Number of participants alive one year post transplant
Time Frame: From treatment start date to death, assessed up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Tagraxofusp-erzs)
Number analyzed (Participants) | 3
Participants | 2

ADVERSE EVENTS:
Time Frame: up to a year post transplant
Arm/Group | Treatment (Tagraxofusp-erzs)
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Tagraxofusp-erzs) (N=3)
Elevated Transaminases (Investigations) | 1 (1)

LIMITATIONS AND CAVEATS:
The protocol was terminated early due to slow participant accrual and the sponsor not willing to provide the study drug.

Stemline is the funder, not the sponsor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-29): https://cdn.clinicaltrials.gov/large-docs/81/NCT04317781/Prot_SAP_000.pdf